CLINICAL TRIAL: NCT07196995
Title: Prospective Multicenter Validation of Whole Body PET/CT Foundation Model for Bone Lesion Detection
Brief Title: Validation of Whole Body PET/CT Foundation Model
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, Principal Investigator, Shanghai 6th People's Hospital
Other Study IDs: PET/CT MODEL 01
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group PET/CT: Whole body PET/CT foundation model
- Group CT: Whole body CT foundation model

SUMMARY:
Prospective multicenter study to validate the diagnostic performance of whole body PET/CT foundation model for bone lesion detection

ELIGIBILITY:
Inclusion Criteria:

* With suspicious lesion in the bone or with elevated serum tumor markers or patient insist
* Over 18 years

Exclusion Criteria:

* Active infection at or adjacent to the puncture site
* Severe coagulation disorders that cannot be corrected
* Random blood glucose > 11.1 mmol/L
* Refuse for pathological confirmation or follow-up
* Extremely debilitated patients or those unable to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: With suspicious lesion in the bone
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance (benign or malignant) | At diagnosis time
  Patient based bone lesion diagnostic performance (benign or malignant)

SECONDARY OUTCOMES:
Diagnostic performance (primary or metastases) | At diagnosis time
  Patient based bone lesion diagnostic performance (primary or metastases)
Pathology prediction | At diagnosis time
  Pathology prediction
Gene prediction | At diagnosis time
  Gene prediction
Prognosis prediction | At diagnosis time
  Prognosis prediction